CLINICAL TRIAL: NCT03459300
Title: Importance of Sleep Deprivation in Differential Diagnosis of Primary Hypersomnia in Reference Centers Rare Hypersomnia
Brief Title: Importance of Sleep Deprivation in Differential Diagnosis of Primary Hypersomnia (Actisom dépistage)
Acronym: Actisom
Status: Completed | Type: Observational
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Other Study IDs: 16047
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Hypersomnia
Keywords: actimetry
MeSH Terms: conditions — Disorders of Excessive Somnolence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
7 to 14 days actimetry recording in order to exclude sleep deprivation just before hospitalisation for differential diagnosis of hypersomnia

DETAILED DESCRIPTION:
This is an observational study

Urine drug screening will also be performe

The suty includes four centers in France

The study duration is of one year

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged > 18 years
* Patient with a sleepiness evoking a primary hypersomnia
* Epworth sleepiness scale > 10
* Information note signed

Exclusion Criteria:

* Patient with type 1 or 2 narcolepsy and/or known hypersomnia
* Frank cataplexy
* Not stable metabolic, neurological or psychiatric disease
* Patient treated by a medicine acting on the central nervous system
* Patient having a shift work or having made a transmeridian flight of more than 3 hours lag in the previous month the research
* Non affiliation to social security
* Pregnancy
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a sleepiness evoking a primary hypersomnia
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
mean total sleep time | 7-14 days before hospitalisation
  mean total sleep time as measured by actimetry durind the 7 - 14 days before hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Maria Antonia QUERA SALVA, MDPhD, Principal Investigator — APHP
Locations (1):
- Hôpital raymond Poincaré, Garches, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No